CLINICAL TRIAL: NCT02986282
Title: Ankle - Brachial Index Measurement in Patients With Atrial Fibrillation Before and After Electrical Cardioversion
Brief Title: Ankle - Brachial Index Measurement in Atrial Fibrillation
Acronym: AFABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Maciej Sinski, M.D., Ph.D., Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AFABI
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation Fluttering
Keywords: ankle - brachial index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Interventions - repeated ankle - brachial index measurement before and after electrical cardioversion in patients with atrial fibrillation
  Interventions: Device: ABI measurement using both doppler and oscillometric method

INTERVENTIONS:
Device: ABI measurement using both doppler and oscillometric method
  Other Names: doppler method (Echo Sounder ES-101EX, Hadeco, Japan and Minimus II, Rister, Germany); oscillometric method (Microlife WatchBP AG, Widnau, Switzerland)

SUMMARY:
Consecutive patients with atrial fibrillation will be admitted to the hospital for electrical cardioversion. Ankle brachial index will be measured three times with oscillometric method and three times with doppler method. Two study sessions will be performed: the first before and the second after electrical cardioversion. The first session will be ended before anesthesia. The second session will be started before a conscious patient will be transported from intensive care unit to general ward.

All the measurements will be taken in the intensive care unit at an ambient temperature of 21° C, after patients will give their written informed consent to participate in the study. All patients will be awake, fasting and in the supine position. ABI will be measured according to the guidelines issued by AHA. Systolic blood pressure will be measured using a Doppler device (Echo Sounder ES-101EX, Hadeco, Japan) and a validated and calibrated aneroid sphygmomanometer (Minimus II, Rister, Germany). Measurement of ABI using oscillometric method will be performed using WatchBP Office ABI system (Microlife WatchBP AG, Widnau, Switzerland). The appropriate cuff size will be used with the width of the cuff being at least 40% of the limb circumference. The arm with higher systolic blood pressure will be used to calculate the ABI. Higher systolic blood pressure measured on the posterior tibial or dorsalis pedis artery will be used to calculate the ABI. During both study sessions ABI measurements will be repeated 3 times with each method in the reverse order of the preceding measurement e.g., in the case of the initial counterclockwise sequence: right arm, right popliteal, right dorsalis pedis, left popliteal, left dorsalis pedis, left arm, right arm, the clockwise sequence will be used, starting and ending with the left arm. The same sequence of limb pressure measurements will be used used during the study.

A sample size calculation was based on the preliminary observations made by the study team. It was calculated that the study sample size of 79 subjects would be needed to detect a difference of 0.1 in the ABI measured in sinus rhythm and during atrial fibrillation, with a two-tailed α of 0.05 and a (1-β) of 0.90. The investigators initial estimate of sample size of 115 patients incorporated an assumption of dropout due to non-effective electrical cardioversion, patient decision to quit study or failure to obtain adequate ABI.

The measurements will be repeated three times with each method and for the each method the mean will be used for the calculations. Investigator - study nurse, trained at the vascular department, will perform all ABI measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing electrical cardioversion due to atrial fibrillation

Exclusion Criteria:

* Circulatory instability
* Use of vasoconstrictive agents
* Limb trauma
* Upper limb artery stenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sinski, M.D., Ph.D., Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be attached to manuscript.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and fifteen consecutive patients with atrial fibrillation admitted to Department of Internal Medicine, Hypertension and Vascular Diseases, Medical University of Warsaw for electrical cardioversion were screened. Participants were recruited to the study from October 2012 up to December 2015.
Groups:
- Single Arm: Interventions - repeated ankle - brachial index measurement before and after electrical cardioversion in patients with atrial fibrillation
  ABI measurement using both doppler and oscillometric method
Period: Overall Study
Arm/Group | Single Arm
Started | 115
Completed | 99
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 99
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 99

OUTCOME MEASURES:

1. Primary Outcome: Difference Between ABI (Ankle - Brachial Index) Before Electrical Cardioversion Using Two Methods (Doppler and Oscillometric).
Description: 3 ABI measurements using both methods (doppler and oscillometric) were performed per participant and the Mean value was considered for each participant, and then a Median value was calculated across participants.
Time Frame: Through the study
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Single Arm
Number analyzed (Participants) | 99
ratio
  ABI oscillometric before | 1.21 [1.13 to 1.27]
  ABI oscillometric after | 1.215 [1.140 to 1.260]
  ABI doppler before | 1.14 [1.0700 to 1.2175]
  ABI doppler after | 1.18 [1.09 to 1.25]
Statistical Analysis 1: Comparison: Single Arm; It was calculated that the study sample size of 79 subjects would be needed to detect a difference of 0.1 in the ABI measured in sinus rhythm and during atrial fibrillation, with a two-tailed α of 0.05 and a (1-β) of 0.90. Our initial estimate of sample size of 115 patients incorporated an assumption of dropout. Intra-observer variability was calculated using intra-class correlation coefficient; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.0600326, 95% CI 2-sided [-0.0799661 to -0.0449876]

2. Secondary Outcome: Difference Between ABI Measured Before and After Electrical Cardioversion Using Doppler Method.
Description: 3 ABI measurements using doppler method were performed per participant and the Mean value was considered for each participant, and then a Median value was calculated across participants
Time Frame: Through the study period
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Single Arm
Number analyzed (Participants) | 99
ratio
  ABI doppler before | 1.14 [1.0700 to 1.2175]
  ABI doppler after | 1.18 [1.09 to 1.25]
Statistical Analysis 1: Comparison: Single Arm; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.0249837, 95% CI 2-sided [-0.039992 to -0.0100226]

ADVERSE EVENTS:
Time Frame: October 2012 - December 2015
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No